CLINICAL TRIAL: NCT06386406
Title: A Mono-centric Clinical Investigation to Evaluate Performance of a Pre-confectioned Plantar Insole for the Treatment of Plantar Heel Pain.
Brief Title: This is a Study to Evaluate a Pre-confectioned Plantar Insole for the Treatment of Plantar Heel Pain
Acronym: TAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORL-ORT-040
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAP insole (Experimental)
  Interventions: Device: TAP insole

INTERVENTIONS:
Device: TAP insole — The patients will have to wear the TAP insole when walking during the everyday life activities.
  This plantar insole is not a custom-made insole but a pre-confectioned one because designed according to two parameters: shoe size and gender.

SUMMARY:
Patients affected by plantar heel pain will be asked to use a pre-confectioned plantar insole for one year.

The aim of the study is to assess if the insole under study allows the patient to reach a better mobility and a faster return to the normal everyday life.

ELIGIBILITY:
Inclusion Criteria:

Male and female adults

* Age ranging 18 to 70 years
* Patients with a history of at least 6 months of plantar fasciitis resistant to other conventional therapies
* Willingness and ability to participate in the trial
* Informed Consent signed by the subject

Exclusion Criteria:

* Diabetes mellitus not controlled pharmacologically
* Rheumatoid arthritis
* Previous foot surgery
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, general physical problem of the participant, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity according to visual analog scale | 3 months
  The pain visual analog scale (VAS) is a validated, self-assessment scale in which patients rate their pain by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The pain VAS will be administered at baseline by the patient himself and at follow-ups.
  A negative change from baseline will indicate an improvement in VAS score and, therefore, in local pain.

SECONDARY OUTCOMES:
Change in pain severity according to visual analog scale | 2 weeks, 6 weeks, 6 and 12 months.
  The pain VAS scale is a validated, self-assessment scale in which patients rate their pain by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The pain VAS will be administered at baseline by the patient himself and at follow-ups.
  A negative change from baseline will indicate an improvement in VAS score and, therefore, in local pain.
Subjective functional recovery based on the Foot Function Index (FFI) score [ | baseline, 2 and 6 weeks, and 3, 6, and 12 months
  Foot function Index measures the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales. The patient will answer each question on a scale from 0 (best) to 10 (worst result), that best describes their foot over the past week. The pain subcategory consists of 9 items and measures foot pain in different situations. The disability subcategory consists of 9 items and measures difficulty performing functional activities because of foot problems. The activity limitation subcategory consists of 5 items and measures limitations in activities because of foot problems. Both total and subcategory scores are calculated.
Quality of life and foot general health through the assessment of the Foot Health Status Questionnaire (FHSQ) | baseline, 2 and 6 weeks, and 3, 6, and 12 months follow-up
  The Foot Health Status Questionnaire (FHSQ) is a self-assessment and trustworthy instrument about health quality regarding specific foot health, initially developed to assess the results of surgical treatment of common foot diseases. It is made of questions regarding foot health and its impact on quality of life. There are 4 subscales: foot pain (4 questions), foot function (4 questions), footwear (3 questions), and general foot health (2 questions). For the subscales of pain, function, and general foot health, there is a 5-point Likert scale of no problems, pain, or limitations to severe problems, pain, or limitations. Responses to footwear questions are on a 5-point bipolar Likert scale from strongly disagree to strongly agree for statements regarding shoe fit, discomfort wearing shoes, and shoe wear available.
Patient satisfaction on a 0-10 numeric rating scale (NRS) | 2 weeks, 6 weeks,3, 6, and 12 months
  self-assessment scale in which patients rate their satisfaction by making a handwritten mark from the lowest satisfaction (0 point) to the highest satisfaction (10 points)

CONTACTS AND LOCATIONS:
Locations (1):
- EOC, Lugano, Switzerland